CLINICAL TRIAL: NCT05542212
Title: The Validity of Intra-cortical Inhibition as a Biomarker of Cognitive Deficits in Schizophrenia and in Predicting the Efficacy of TMS Treatment
Brief Title: Intra-cortical Inhibition and Cognitive Deficits in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Weiqing Liu, Associate Professor, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDJWLL-2021028
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMS treatment group (Experimental): 1. Receive ICI test and MATRICS test.
  2. Receive active iTBS treatment on the dlPFC for 4 weeks, 1 treatment a day and 5 days a week.
  Interventions: Device: Transcranial Magenetic Stimulation
- TMS Sham Control Group (Sham Comparator): 1. Receive ICI test and MATRICS test.
  2. Receive sham TMS treatment on the dlPFC for 4 weeks, 1 treatment a day and 5 days a week.
  Interventions: Device: Sham Transcranial Magenetic Stimulation
- Normal Control (No Intervention): 1. Receive ICI test and MATRICS test.

INTERVENTIONS:
Device: Transcranial Magenetic Stimulation — Intermittent Theta Burst Stimulation (iTBS) treatment plan: iTBS treatment for the left dlPFC were used for a total of 20 treatments (one time each Monday to Friday, continuous treatment for 4 weeks).
  Arms: TMS treatment group
Device: Sham Transcranial Magenetic Stimulation — Sham stimulation: The coil angle is set at 90° to the scalp for Sham stimulation of the left dlPFC for a total of 20 treatments (one time each Monday to Friday, continuous treatment for 4 weeks).
  Arms: TMS Sham Control Group

SUMMARY:
Cognitive deficit is a core symptom of schizophrenia (SZ), but its pathological mechanism is poorly understood and the treatment effect is poor. The excitatory-inhibitory microcircuit (E-I) function imbalance formed by inhibitory interneurons and excitatory pyramidal cells in the cerebral cortex is a new mechanism of cognitive deficits in SZ discovered in recent years. Cortical E-I is expected to be a new target for the treatment of cognitive deficits in SZ. Paired transcranial magnetic stimulation (ppTMS)-induced intracortical inhibition (ICI) is dependent on cortical E-I functional integrity. We found that ICI deficiency is stable in SZ and is closely related to cognitive function. Therefore, ICI is likely to be a system-level biomarker for cognitive deficits caused by E-I imbalance. However, no study has yet explored the genetic basis of ICI and its impact on the occurrence, development and treatment response of cognitive deficits in SZ. Based on this, we intend to verify the value of ppTMS-induced ICI as a biomarker of E-I imbalance in SZ patients and normal controls at different stages: 1. To explore the correlation of ICI with multidimensional cognitive deficits and E-I pathway genes; 2. To explore ICI Combining candidate genes and serum inflammatory factors can predict whether TMS can improve the efficacy of cognitive deficits, and can be used for precise treatment of SZ cognitive deficits at the level of pathological mechanisms.

DETAILED DESCRIPTION:
Study 1. In schizophrenia patients at different stages and normal controls, ppTMS-induced M1 intracortical inhibition was used as a candidate biomarker to comprehensively analyze its correlation with cognitive deficits in the seven dimensions of schizophrenia;

1. To compare the differences in ppTMS-induced intracortical inhibition (SICI and LICI) in the M1 area between schizophrenic patients in the first drug-free period and remission period, and between patients and normal controls;
2. To compare the differences in the 7 cognitive function dimensions of the MCCB between schizophrenic patients in the first episode of drug-free period and remission period, and between patients and normal controls;
3. Analyze the correlation between intracortical inhibition (SICI and LICI) and seven cognitive function dimensions in first-episode drug-free schizophrenia, remission schizophrenia, and normal controls.

Study 2. In patients with schizophrenia and normal controls, to investigate whether there is a correlation between ppTMS-induced intracortical suppression in the M1 area and susceptibility genes that can regulate the function of the E-I microcircuit;

1. Compare the 12 susceptibility genes related to the functional regulation of the E-I microcircuit between patients with schizophrenia and normal controls (including: GABA receptor encoding genes of different subtypes, NMDA receptor encoding genes and others that may affect E-I The distribution difference of 23 single nucleotide polymorphism sites (SNP) in the candidate genes of microcirculation and cognitive function) between the two groups;
2. Compare the effects of the genotypes of each SNP site and the haplotypes of each SNP on the intracortical inhibitory indicators (SICI and LICI) of schizophrenia in the above samples;
3. Further analyze whether the SNP sites found in the previous part that have a significant impact on SICI and LICI also affect cognitive functions in certain dimensions in the above samples. And analyze the potential causal relationship between susceptibility genes and intracortical inhibitory indicators and cognitive deficits;

Study 3. Intermittent theta-burst transcranial magnetic stimulation (iTBS) or sham stimulation intervention on the left dlPFC in patients with schizophrenia, analysis of the efficacy of iTBS in improving cognition and intracortical inhibition indicators at baseline and during the treatment interval and treatment The relationship between post-variation and E-I microcircuit function-related susceptibility genes and intracortical inhibition to predict the cognitive efficacy of iTBS.

1. To analyze whether iTBS treatment can effectively reverse the cognitive deficits in patients with first-episode drug-free and remission schizophrenia;
2. To further analyze whether iTBS treatment can reverse the intracortical inhibitory deficits in patients with first-episode drug-free and remission schizophrenia;
3. Analyze whether the efficacy of iTBS in improving cognitive deficits is related to pre-treatment intracortical inhibition (SICI and LICI) in first-episode drug-free and remission schizophrenia patients; and whether the efficacy of iTBS is related to treatment interval and treatment The magnitude of the change in intracortical inhibition after the end correlates;
4. Establish a predictive model for the early prediction of the efficacy of iTBS in improving cognitive deficits by E-I microcircuit function regulation susceptibility gene SNP and SICI and LICI indicators.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers or Schizophrenia patients: To be diagnosed as "schizophrenia" by the research doctor using the DSM-IV-TR Axis I Disorder Clinical Examination Guidelines Research Edition (SCID-I/P) ;
* Right-handed;
* Education level of junior high school or above;
* The patient is a permanent resident of Shanghai, and there is no plan to move to another place in the next 3 months, and can cooperate with follow-ups;
* Has signed an informed Consent;
* The patient should meet one of the following two conditions: A. First-time onset of schizophrenia, never taking antipsychotics, and PANSS score ≥ 70 points; B. Schizophrenia with less than 3 episodes Symptomatic patients, whose symptoms were relieved within the past 3 months (PANSS score <60 points).

Exclusion Criteria:

* Those who have local or diffuse brain injury or severe brain trauma, and those who have intracranial hypertension;
* Those who have a history of epileptic seizures or a family history of idiopathic epilepsy;
* Those who have paramagnetic or non-paramagnetic metals in the head and neck Implants (such as cochlear implants, titanium clips, etc.);
* Those who have Alcohol dependence and other drug abusers;
* Those who have Severe heart disease, pacemaker or stent implantation;
* Have taken benzodiazepines or received TMS or electroconvulsive therapy within 3 months;
* Patients with moderate or higher depression (HAMD≥17) and anxiety (HAMA≥14) mood;
* Those who are considered unsuitable for enrollment by the researchers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline Speed of Information Processing score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by summation of Trail Making Test, BACS Symbol coding and Verbal Fluency scores in MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia)
Percent Change from Attention/Vigilance score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by Continuous Performence Test scores in MATRICS
Percent Change from Working Memory score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by WMS-III SS scores in MATRICS
Percent Change from Verbal Learning score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by HVLT-R scores in MATRICS
Percent Change from Visual Learning score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by BVMT-R scores in MATRICS
Percent Change from Reasoning and Problem Solving score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by NAB Mazes scores in MATRICS
Percent Change from Social Cognition score at 2 weeks and 4 weeks assessed by MATRICS toolkit. | Baseline, 2 weeks, 4 weeks
  Measured by MSCEIT Branch 4 scores in MATRICS

SECONDARY OUTCOMES:
Change from baseline Intracortical inhibition | Baseline, 2 weeks, 4 weeks
  Intracortical inhibition is the Percent Inhibition of Movement Evokded Potentials of the test TMS stimulus by a conditinal TMS stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Liu, Ph.D, Principal Investigator — Shanghai Pudong New Area Mental Health Center
Locations (1):
- Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No